CLINICAL TRIAL: NCT05414747
Title: A Prospective Multi-Site Open Label Randomized Controlled Clinical Investigation of the Safety and Effectiveness of the ABV-1701 Ocular Endotamponade (OE)
Brief Title: Clinical Investigation of the Safety and Effectiveness of the ABV-1701 Ocular Endotamponade (OE)
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: waiting the new batch of investigational product.
Sponsor: BioFirst Corporation (Industry)
Collaborators: ABVC BioPharma, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABV-1701-02
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Retinal Detachment
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Intervention Model Description: ABV-1701 Ocular Endotamponade
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants randomized to ABV-1701 Ocular Endotamponade (Experimental): Participants randomized to the interventional device ABV-1701 Ocular Endotamponade undergoing the vitrectomy surgery for uncomplicated retinal detachment
  Interventions: Device: ABV-1701
- Participants randomized to SF6 Gas Ocular Endotamponade (Active Comparator): Participants randomized to the control device SF6 Gas Ocular Endotamponade undergoing the vitrectomy surgery for uncomplicated retinal detachment
  Interventions: Device: SF6 Gas

INTERVENTIONS:
Device: ABV-1701 — ABV-1701 is an injectable, in-situ-forming hydrogel, composed of oxidized hyaluronic acid (oxi-HA) and adipic acid dihydrazide (ADH)
  Arms: Participants randomized to ABV-1701 Ocular Endotamponade
Device: SF6 Gas — SF6 is a commercial gas tamponade as a vitreous substitute in pars-plana vitrectomy surgery (PPV)
  Arms: Participants randomized to SF6 Gas Ocular Endotamponade

SUMMARY:
A Prospective Multi-Site Open Label Randomized Controlled Clinical Investigation of the Safety and Effectiveness of the ABV-1701 Ocular Endotamponade (OE)

DETAILED DESCRIPTION:
A Prospective Multi-Site Open Label Randomized Controlled Clinical Investigation of the Safety and Effectiveness of the ABV-1701 Ocular Endotamponade (OE) The objective of the investigation is to document the safety and effectiveness of the ABV-1701 OE when compared to the SF6 Gas OE.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults aged 18 years or older on the day of screening;
2. Uncomplicated retinal detachment defined as one of the following:

   1. The first instance of a small macular hole (<400 microns)
   2. The first instance of a single small (<400 microns) primary tear extending less than 2 clock hours. There is no limit on the number or the position of the break(s). The tear can be PVR grade A (Vitreous haze and pigment clumps) or B (Surface retinal wrinkling, rolled edges of the retinal, retinal stiffness, and vessel tortuosity), but not more than grade B
3. Scheduled vitrectomy with vitreous substitute;
4. Must be able and willing to provide written informed consent, attend all scheduled visits and comply with all study procedures;

Exclusion Criteria:

1. Any active intraocular or periocular infection or inflammation;
2. Vitreous haemorrhage
3. Complicated Retinal detachments due to the following:

   1. Detachment due to Trauma
   2. Detachment due to Uveitis
   3. Chronic detachments defined as 2 or more surgeries
   4. PVR grade CA
4. Only one functional eye;
5. Ocular disorders in the study eye that could confound the interpretation of the study results. i.e. macular edema not requiring vitrectomy surgery, choroidal neovascularization;
6. High refractive error demonstrating >6 diopters of myopia;
7. An ophthalmic condition that reduces the clarity of the ocular media that may interfere with ophthalmic examination or imaging. i.e. Cataract, corneal opacity;
8. Uncontrolled glaucoma defined as intraocular pressure >30 mmHg on maximal therapy;
9. Aphakia or the absence of the posterior capsule;
10. Known hypersensitivity to hyaluronic acid or acid dihydrazide (ADH);
11. Uncontrolled blood pressure defined as systolic value >160 mmHg or diastolic value > 100 mmHg at screening;
12. Uncontrolled diabetes defined as glycated hemoglobin (HbA1c) >12%;
13. Pregnant or breastfeeding at the time of screening;
14. Women of childbearing potential, defined as women physiologically capable of becoming pregnant unless using effective methods of contraception during the study period. The effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the participant). Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) is not acceptable.
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
    * Male sterilization (at least 6 months prior to screening). For female participants on the study, the vasectomized male partner should be the sole partner for that participant.
    * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps).
    * Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
    * Placement of an intrauterine device (IUD) or intrauterine system (IUS).
15. Participation in any study involving an investigational drug or device within the past 30 days or ongoing participation in a study with an investigational drug or device.
16. Any clinical evidence that the investigator feels would place the participant at increased risk with the investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Rate of anatomical retinal attachment success | 90 days
  Rate of anatomical retinal attachment success (percent) at Day 90 from an uncomplicated retinal detachment at baseline. Successful cases measured by the absence of any adverse event or complication at Day 90.

SECONDARY OUTCOMES:
Change in best-corrected visual acuity (BCVA) | 180 days
  Change in best-corrected visual acuity (BCVA) from baseline
Number of surgeries | 90 days
  Number of surgeries (required to reattach the retina if recurrent retinal detachment occurs) between Day 0 and Day 90
Secondary surgical/medical interventions - IOP elevation | 180 days
  Number of secondary surgical/medical interventions due to IOP elevation
Secondary surgical/medical interventions - cataract formation | 180 days
  Number of secondary surgical/medical interventions due to cataract formation
Secondary surgical/medical interventions - corneal abnormalities | 180 days
  Number of secondary surgical/medical interventions due to corneal abnormalities
Secondary surgical/medical interventions - adverse events | 180 days
  Number of secondary surgical/medical interventions due to adverse events (AE)s

CONTACTS AND LOCATIONS:
Overall Officials: Richard CH King, Ph.D., Study Director — ABVC BioPharma, Inc
Locations (4):
- Australia (2):
  - Sydney Eye Hospital, Sydney, New South Wales
  - East Melbourne Eye Group, Melbourne, Victoria
- Thailand (2):
  - Ramathibodi Hospital, Bangkok
  - Srinagarind Hospital, Khon Kaen

IPD SHARING:
Plan to Share IPD: No